CLINICAL TRIAL: NCT04788355
Title: Hydroxychloroquine and Apixaban: Analysis of Physiological Parameters for the Prevention of Complications in Patients With Infection With the New Coronavirus (Covid-19). A Randomized Clinical Trial
Brief Title: Prevention of Complications (SARS-CoV-2): Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Collaborators: Pfizer (Industry); Apsen Farmaceutica S.A. (Industry); Dermadia (Unknown); Methodos Laboratory (Unknown); Biofarma (Industry)
Responsible Party: Principal Investigator, José Dias da Silva Neto, Doctor, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HA and A COVID 19
Record Dates: First submitted 2020-09-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Complication
Keywords: Complications; Novel coronavirus 2019; SARS-CoV-2; Chloroquine; Anticoagulants
MeSH Terms: interventions — Control Groups; apixaban; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Clinical study that will evaluate the action of drugs combined or not to reduce complications of patients with covid 19
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will not know which groups the patients belong to
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group standard treatment (Active Comparator): Patients will be treated only with standard hospital treatment
  Interventions: Drug: Control group (standard hospital treatment)
- Group Hydroxychloroquine (Experimental): Patients will be treated with Hydroxychloroquine associated with standard hospital treatment
  Interventions: Drug: Control group (standard hospital treatment); Drug: Group Hydroxychloroquine
- Group Hydroxychloroquine e Apixaban (Experimental): Patients will be treated with Hydroxychloroquine associated with apixaban and standard hospital treatment
  Interventions: Drug: Control group (standard hospital treatment); Drug: Group Hydroxychloroquine and apixaban
- Group Apixabana (Experimental): Patients will be treated with apixaban associated with standard hospital treatment
  Interventions: Drug: Control group (standard hospital treatment); Drug: Group Apixaban

INTERVENTIONS:
Drug: Control group (standard hospital treatment) — Medications defined by the hospital involved in the study
  Other Names: Drug protocols recommended by WHO and the Ministry of Health that make up the standard hospital treatment
Drug: Group Hydroxychloroquine — Patients in this group will receive hydroxychloroquine orally 200 mg every 12 hours for 7 days. In addition, patients in this group will receive standard medication for COVID-19 which is part of the hospital protocol involved in the study.
  Other Names: Hydroxychloroquine associated with standard treatment of the hospital involved in the study
  Arms: Group Hydroxychloroquine
Drug: Group Hydroxychloroquine and apixaban — Patients in this group will receive hydroxychloroquine orally 200 mg every 12 hours for 7 days + apixaban orally 2.5 mg every 12 hours, also for 14 days (prophylactic dose). In addition, patients in this group will receive standard medication, which is the protocol of the hospital involved in the study.
  Other Names: Hydroxychloroquine, Apixaban and standard treatment
  Arms: Group Hydroxychloroquine e Apixaban
Drug: Group Apixaban — Patients in this group will receive apixaban 2.5 mg orally every 12 hours, also for 14 days (prophylactic dose). In addition, patients in this group will receive standard medication, which is the protocol of the hospital involved in the study.
  Other Names: Apixaban and standard treatment
  Arms: Group Apixabana

SUMMARY:
Viral diseases have always posed a threat to public health. Recently, the SARS-Cov2 virus spread in an epidemic that began in China and soon spread globally, making its study extremely relevant, in order to seek mechanisms to combat it. Therefore, this study seeks to evaluate the benefit of using Hydroxychloroquine with or without Apixaban in the early treatment of patients with suspected COVID-19. Prospective, randomized, double-blind, controlled study, performed at Hospital das Clínicas Samuel Libânio (Universidade do Vale do Sapucaí) UNIVÁS, Pouso Alegre, Minas Gerais, Brasil. Patients treated in the emergency department who are reported as suspected cases of COVID-19 patients will be included, according to current guidelines. Will be randomized into 4 groups: Hydroxychloroquine, Hydroxychloroquine + Apixabana, only Apixabana and Control group, all receiving standard treatment recommended. Included patients will be monitored during hospitalization or remotely assisted in home treatment. Clinical, laboratory, electrocardiographic and image evaluation criteria will be considered to assess the evolution in 7 and 14 days after inclusion. Results will be subjected to appropriate statistical analysis, with sample calculation. An early therapeutic approach is proposed in suspected and confirmed patients with COVID-19, with the hope of reducing hospitalizations and severe forms of the disease.

DETAILED DESCRIPTION:
The early administration of HCQ or in association with apixaban, could prevent worsening of suspected COVID-19, as well as preventing hospitalizations and the need for intensive treatment. In patients with mild to moderate disease, the use of hydroxychloroquine or hydroxychloroquine with apixaban or apixaban alone, could be able to reduce disease progression on an ordinal scale of outcome (including use of mechanical ventilation and death) and decrease the likelihood of hospitalization or worsening of clinical conditions.

ELIGIBILITY:
Inclusion criteria:

* Patients with suspected or confirmed covid-19, above 18 years old
* Patients with time between symptom onset and inclusion ≤ 14 days
* Patients with time between hospital stay and inclusion ≤ 48 hours

Exclusion criteria:

* Patients tested negative for covid-19 by rt-pcr, serological or rapid test method
* Patients unable to swallow for any reason
* Patients with an extended qt interval, defined as a corrected qt (qtc) for heart rate above 450 ms for men and 470 ms for women
* Patients with liver toxicity, defined as ast / alt or increased bilirubin
* Patients with ventricular arrhythmias
* Patients with bleeding, major hematoma or blood dyscrasia;
* Patients who, at any time during the process, choose to give up participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Patients in home isolation will be followed for (telemedicine) 14 days. The Beck scale will assess anxiety. Questions will be asked to patients about their health conditions. The answers will be tabulated in a spreadsheet composed of the following result | 14 evaluation days after inclusion in the study
  The Beck scale will assess anxiety. Questions asked by telemedicine: cough, dyspnea, fatigue, malaise, myalgia, runny nose, odynophagia, anosmia, ageusia, headache, anorexia, abdominal pain, conjunctival congestion, diarrhea, nausea, vomiting, palpitation, bleeding, atypical symptoms. The parameters for such telemedicine evaluations were: yes or no.

SECONDARY OUTCOMES:
Assessment of the presence or absence of secondary complications for patients in home isolation or hospitalized, after using the drugs. | 14 evaluation days after inclusion in the study
  The relationship between the use of medications in the initial interventions and the presence or absence of secondary complications will be assessed both for patients in home isolation and for hospitalized patients. As for patients who are hospitalized, the following topics will be included in the table: use of oxygen therapy, mechanical ventilation, death. The parameters for answers will be yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Univás, Pouso Alegre, Minas Gerais, Brazil